CLINICAL TRIAL: NCT00846781
Title: Study 08-114 Open-label Extension of Study 08-110 - A Multi-Center Study of Denufosol Tetrasodium Inhalation Solution in Patients With Cystic Fibrosis Lung Disease (P08642)
Acronym: DEFY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P08642; 08-114
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Denufosol tetrasodium Inhalation Solution (Experimental)
  Interventions: Drug: Denufosol tetrasodium Inhalation Solution

INTERVENTIONS:
Drug: Denufosol tetrasodium Inhalation Solution — 60 mg by oral inhalation three times daily

SUMMARY:
The purpose of this study is to obtain data on the potential of long-term treatment with denufosol to improve the clinical course of CF lung disease in patients with mildly impaired lung function and to provide CF patients who completed study 08-110 continued access to denufosol.

ELIGIBILITY:
Inclusion Criteria:

* Completed Study 08-110

Exclusion Criteria:

* A female patient will not be eligible for the study if she is of childbearing potential and is pregnant, lactating, and/or not practicing an acceptable method of birth control (e.g., abstinence, hormonal or barrier methods, partner sterilization, or intrauterine device).
* Have a condition that might affect compliance with study procedures

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Rate of change in lung function, as measured by change in FEV1 | 160 Weeks

SECONDARY OUTCOMES:
Change in absolute FEV1 from baseline | Weeks 12, 24, 36, 48, 72, 96, 120, 144, and 160
Change in FEV1 percent predicted value from baseline | Weeks 12, 24, 36, 48, 72, 96, 120, 144, and 160
Change in FEF25%-75% and forced vital capacity (FVC) from baseline | Weeks 12, 24, 36, 48, 72, 96, 120, 144, and 160
Incidence of pulmonary exacerbations | 160 Weeks
Changes in Pseudomonas aeruginosa status | 160 Weeks
Number of days of intravenous (IV) antibiotic use for a respiratory complaint | 160 Weeks
Incidence of hospitalizations/Emergency room (ER) visits for a respiratory complaint | 160 Weeks
Number of days hospitalized for a respiratory complaint | 160 Weeks
Incidence of treatment emergent adverse events (AEs), serious adverse events (SAEs) and withdrawals due to AEs | 160 Weeks
Incidence of patients with significant decrease in absolute FEV1 at any visit from baseline | 160 Weeks
Changes in physical exam findings including height, weight, and body mass index from baseline | Weeks 48, 96, and 160
Changes in hematology, serum chemistry, and urinalysis parameters from baseline | Weeks 24, 48, 72, 96, 120, 144, and 160
Incidence of hospitalizations/ER visits | 160 Weeks
Incidence of early discontinuations from the study | 160 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Smiley, MD, Study Director — Medical Monitor